CLINICAL TRIAL: NCT02641093
Title: Phase II Investigation of Adjuvant Combined Cisplatin and Radiation With Pembrolizumab in Resected Head and Neck Squamous Cell Carcinoma
Brief Title: Phase II Trial of Adjuvant Cisplatin and Radiation With Pembrolizumab in Resected Head and Neck Squamous Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Trisha Wise-Draper (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Trisha Wise-Draper, Principal Investigator, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCCI-HN-15-01
Record Dates: First submitted 2015-12-21; First posted 2015-12-29 (Estimated); Results first posted 2023-05-06 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — pembrolizumab; Surgical Procedures, Operative; Radiotherapy; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pembrolizumab (Experimental): Pembrolizumab in combination with standard of care surgery followed by radiation therapy with or without cisplatin
  Interventions: Drug: Pembrolizumab; Procedure: Surgery; Radiation: Radiation Therapy; Drug: Cisplatin

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab administered one week prior to surgery and then every three weeks in the adjuvant setting for a total of 7 doses.
  Other Names: Keytruda
Procedure: Surgery — gross total surgical resection
Radiation: Radiation Therapy — 60-66 Gy over 6 weeks
Drug: Cisplatin — Weekly during radiation therapy for 6 doses only for patients with high risk pathological features

SUMMARY:
The purpose of this research study is to test the safety and the benefit of adding pembrolizumab (a therapy that activates the immune system to fight cancer) to standard of care treatment for head and neck cancer. The standard of care treatment will include surgery followed by radiation for 6 weeks. Some patients may also receive cisplatin as standard of care once a week for 6 weeks if the cancer is found to be "high risk". High risk includes cancer that was not completely removed (positive margins) or cancer that has invaded through the outer lining of your lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for resection with one or more of the following

  1. Any T stage with ≥ N2 disease;
  2. T4 disease, any N stage;
  3. T3 Oral Cavity, any N stage; or
  4. Clinical evidence of extra-capsular extension on scans.
* Must be willing to undergo definitive resection with neck dissection.
* Performance status 0 or 1 on Eastern Cooperative Oncology Group Performance Scale.
* Adequate labs
* Appropriate staging imaging.

Exclusion Criteria:

* Diagnosis of immunodeficiency or receiving systemic steroid therapy or immunosuppressive therapy within 7 days prior to planned first dose of trial treatment.
* Nasopharyngeal or sinonasal carcinoma
* Confirmed metastatic disease
* Human Papillomavirus (HPV)+ disease of the oropharynx
* Known history of active tuberculosis (TB), autoimmune disease, pneumonitis, infection, HIV, Hepatitis B, or Hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2025-11-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Trisha Wise-Draper, MD, PhD, Principal Investigator — University of Cincinnati
Locations (6):
- United States (6):
  - University of Louisville - James Graham Brown Cancer Center, Louisville, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - MD Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab: * Pembrolizumab in combination with standard of care surgery followed by radiation therapy with or without cisplatin.
  * Pembrolizumab: Pembrolizumab administered intravenously one week prior to surgery and then every three weeks in the adjuvant setting for a total of 7 doses. The dose is 200 mg every three weeks.
  * Surgery: gross total surgical resection
  * Radiation Therapy: 60-66 Gy over 6 weeks
  * Cisplatin: administered intravenously at 40 mg/m2 weekly during radiation therapy for 6 doses only for patients with high-risk pathological features
Period: Overall Study
Arm/Group | Pembrolizumab
Started | 96
Completed | 67
Not Completed | 29

BASELINE CHARACTERISTICS:
Population: This is the total number of subjects. Other sections report different subject numbers as they are subsets of 92.
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 92
Age, Continuous [Median (Full Range); unit: years] | 59 [27 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 87
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Related Adverse Effects
Description: Number of participants with treatment related adverse effects as assessed using CTCAE v4.0 of pembrolizumab when combined with radiation alone and chemoradiation. Compared as percentage of grade 3 and 4 adverse events with historical control percentages.
Time Frame: All adverse events were recorded from the time the consent form is signed through 30 days following cessation of treatment. Any AE related to study drug after 30 days post treatment, subjects were followed until resolution.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 92
Participants | 78

2. Primary Outcome: Disease Free Survival in Resected High Risk Patients Treated With Adjuvant Pembrolizumab and Chemoradiation
Description: • High risk is defined as those with biopsies that have the following features: extracapsular spread or those with positive surgical margins.
Time Frame: 1 year
Population: • High risk is defined as those with biopsies that have the following features: extracapsular spread or those with positive surgical margins.
Measure: Number (95% Confidence Interval); unit: percentage of high risk participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 44
percentage of high risk participants | 66 [55 to 84]

3. Primary Outcome: Disease Free Survival in Resected Intermediate Risk Patients Treated With Adjuvant Pembrolizumab and Radiation
Description: • Intermediate risk is defined as those with biopsies that do not have the following features: extracapsular spread or those with positive surgical margins.
Time Frame: 1 year
Population: • Intermediate risk is defined as those with biopsies that do not have the following features: extracapsular spread or those with positive surgical margins.
Measure: Number (95% Confidence Interval); unit: percentage of intermediate participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 31
percentage of intermediate participants | 96 [90 to 100]

4. Secondary Outcome: Tumor Immune Response to Pembrolizumab as Defined by PD-L1 CPS in the Baseline Tumor Tissue
Description: Change in distribution of the tumor immune microenvironment after Pembrolizumab administration in tumor biopsy tissue using markers of T cells and T cell activation using PD-L1 CPS. PD-L1 CPS is defined as the PD-L1 combined positive score. PD-L1 CPS is defined as Combined positivity score (CPS) was calculated by summing the numbers of PD-L1-positive tumor cells and immune cells and dividing by the total number of viable tumor cells. Additionally, PD-L1 is a protein that helps the body immune system remain in control.
  The denominator in this case is 72 subjects that were evaluable. Evaluable means the subject had a pre-surgery pembrolizumab and a biopsy taken. The numerators are explained below.
Time Frame: 1 week between receiving a pre-surgery dose of pembrolizumab and surgery when the biopsy was taken
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 72
Participants
  PD-L1 CPS in Baseline tumor tissue was zero | 20
  PD-L1 CPS in Baseline tumor tissue was ≥1 | 52

5. Secondary Outcome: Overall Survival in Resected Intermediate Risk Patients Treated With Adjuvant Pembrolizumab and Radiation
Description: as for outcome 3
Time Frame: 1 year
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of intermediate participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 31
percentage of intermediate participants | 100 [100 to 100]

6. Secondary Outcome: Overall Survival in Resected High Risk Patients Treated With Adjuvant Pembrolizumab and Chemoradiation
Description: as for outcome 2
Time Frame: 1 year
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of high risk participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 44
percentage of high risk participants | 93 [85 to 100]

ADVERSE EVENTS:
Time Frame: All adverse events were recorded from the time the consent form is signed through 30 days following cessation of treatment. Any AE related to study drug after 30 days post treatment, subjects were followed until resolution, approximately 3.61 months.
Description: Adverse events were reviewed for at all protocol specified timepoints by reviewing medical records, laboratory results and through subject self-report. Adverse events collection occurred from within the intent-to-treat population and therefore was inclusive of more subjects than those determined to be evaluable.
Arm/Group | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 20/96
Serious Adverse Events (participants affected / at risk) | 43/96
Other Adverse Events (participants affected / at risk) | 92/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=96)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Anorectal infection (Infections and infestations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Bone infection (Infections and infestations) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Delirium (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Edema face (General disorders) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (2) — Hematochezia odynophagia
Hematoma (Vascular disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 4 (7) — alpha hemolytic strep left side neck abscess rupture Coagulase-negative staphylococci neck abscesses Multifocal pneumonia Intestinal infection due to Clostridium difficile Infection, right leg graft site
Laryngeal fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Lung infection (Infections and infestations) | 4 (5)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 3 (4) — Failure to thrive
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Neutrophil count decreased (Investigations) | 1 (1)
Pain (General disorders) | 1 (1)
Pancreatitis (Infections and infestations) | 1 (1)
Pharyngeal fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Hypoxemia
Salivary gland infection (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Immune system disorders) | 4 (5)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1) — free flap failure
Syncope (Nervous system disorders) | 1 (1)
Tracheal obstruction (Injury, poisoning and procedural complications) | 1 (1)
Tracheitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2)
Venous injury (Injury, poisoning and procedural complications) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (5)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2)
Wound infection (Infections and infestations) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=96)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 8 (10)
Activated partial thromboplastin time prolonged (Investigations) | 4 (7)
acute kidney injury (Renal and urinary disorders) | 4 (4)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
agitation (Psychiatric disorders) | 3 (3)
Alanine aminotransferase increased (Investigations) | 10 (14)
Alkaline phosphatase increased (Investigations) | 4 (4)
Allergic reaction (Immune system disorders) | 3 (3)
allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
alopecia (Skin and subcutaneous tissue disorders) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 31 (67)
Anorexia (Metabolism and nutrition disorders) | 28 (43)
Anxiety (Psychiatric disorders) | 18 (22)
Aphonia (Nervous system disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 8 (10)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1)
Autoimmune disorder (Immune system disorders) | 1 (1)
Back Pain (General disorders) | 6 (6)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 9 (9) — microcytic anemia Cervical adenopathy low iron and low iron saturation Eosinophilic leukocytosis blood clot
Blood bilirubin increased (Investigations) | 1 (2)
Blurred vision (Eye disorders) | 4 (4)
Bone infection (Infections and infestations) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Burn (Injury, poisoning and procedural complications) | 1 (1)
cardiac disorders other specify (Cardiac disorders) | 1 (1) — heart rate fluctuating between 30's - 100's
CD4 lymphocytes decreased (Investigations) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 2 (2)
Chills (General disorders) | 3 (3)
Chronic kidney disease (Renal and urinary disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1)
Concentration impairment (Nervous system disorders) | 1 (1)
confusion (Psychiatric disorders) | 1 (1)
conjunctivitis (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 41 (49)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (22)
Creatinine increased (Investigations) | 11 (14)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 16 (21)
Delirium (Psychiatric disorders) | 2 (3)
Dental Caries (Gastrointestinal disorders) | 4 (5)
Depression (Psychiatric disorders) | 12 (16)
Dermatitis radiation (Injury, poisoning and procedural complications) | 46 (66)
Diarrhea (Gastrointestinal disorders) | 24 (29)
Dizziness (Nervous system disorders) | 14 (14)
Dry eye (Eye disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 36 (43)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (6)
Duodenal hemorrhage (Gastrointestinal disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 12 (15)
Dysgeusia (Nervous system disorders) | 34 (45)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 56 (97)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 13 (17)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 3 (3) — Ear clogging up and popping Ear popping and bleeding
Ear pain (Ear and labyrinth disorders) | 6 (10)
Edema face (General disorders) | 32 (40)
Edema limbs (General disorders) | 10 (11)
Encephalopathy (Nervous system disorders) | 1 (1)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (1) — Diabetes Mellitus
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 10 (10)
Esophageal pain (Gastrointestinal disorders) | 1 (1)
eye disorders - other, specify (Eye disorders) | 1 (1) — redness on left lower lid
Eyelid function disorder (Eye disorders) | 1 (1)
Facial pain (General disorders) | 7 (7)
Fall (General disorders) | 3 (3)
Fatigue (General disorders) | 64 (75)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Fever (General disorders) | 9 (11)
Fibrinogen decreased (Investigations) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 7 (10)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 34 (35) — unusual sensation R buccal mucosa mouth blisters odynophagia drooling Mouth sores thick secretions Lip blisters irritable bowels bloody stool
General disorders and administration site conditions - Other, specify (General disorders) | 4 (4) — raised lesion R mouth edge of flap decreased activity stoma pain
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (4)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (1)
head soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 11 (12)
Hearing impaired (Ear and labyrinth disorders) | 5 (8)
Heart failure (Cardiac disorders) | 1 (1)
hematoma (Vascular disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 5 (7)
hemorrhoids (Gastrointestinal disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Hepatitis viral (Infections and infestations) | 1 (1)
Vascular disorders - other, specify (Vascular disorders) | 1 (1) — Transient elevated blood pressure
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Hot flashes (Vascular disorders) | 3 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 13 (23)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 8 (19)
Hyperthyroidism (Endocrine disorders) | 6 (6)
Hyperuricemia (Metabolism and nutrition disorders) | 4 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (10)
Hypocalcemia (Metabolism and nutrition disorders) | 6 (10)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 16 (22)
Hypomagnesemia (Metabolism and nutrition disorders) | 18 (22)
Hyponatremia (Metabolism and nutrition disorders) | 12 (23)
Hypoparathyroidism (Endocrine disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 9 (15)
Hypotension (Vascular disorders) | 11 (12)
Hypothyroidism (Endocrine disorders) | 13 (14)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Immune system disorders - Other, specify (Immune system disorders) | 1 (1) — Adenopathy
Infections and infestations - Other, specify (Infections and infestations) | 41 (47) — Thrush, Various drainage Alpha hemolytic Strep & Parvimonas micra Neck infection/abcess mycobacterial abscessus jaw infection C. Difficile methicillin-resistant staphylococcus aureus
Infusion related reaction (General disorders) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 20 (20) — Rotator Cuff Injury Chyle leak accidental trach decannulation pain or bleeding at G-tube site exposed bone in mouth\ Drain fell out fistula lip purulent - drainage buttock wound toe wound False Lumen Surgical flap failure
INR increased (Investigations) | 2 (2)
Insomnia (Psychiatric disorders) | 20 (20)
Investigations - Other, specify (Investigations) | 7 (7) — decreased BUN decreased albumin ketones in urine Cold intolerance Increased BUN
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 3 (3)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2)
lip infection (Infections and infestations) | 1 (1)
Lip pain (Gastrointestinal disorders) | 2 (2)
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 1 (1)
Localized edema (General disorders) | 15 (15)
Lung infection (Infections and infestations) | 2 (2)
Lymphedema (Vascular disorders) | 29 (32)
Lymphocyte count decreased (Investigations) | 11 (39)
Lymphocyte count increased (Investigations) | 1 (1)
memory impairment (Nervous system disorders) | 1 (1)
Meningismus (Nervous system disorders) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 5 (5) — Malnutrition
Movements involuntary (Nervous system disorders) | 1 (1)
Mucosal infection (Infections and infestations) | 8 (9)
Mucositis oral (Gastrointestinal disorders) | 49 (81)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 24 (26) — neck stiffness jaw pain Degenerative disc disease pain at graft site
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Nail infection (Infections and infestations) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 42 (60)
Neck edema (General disorders) | 16 (19)
Neck pain (Musculoskeletal and connective tissue disorders) | 27 (30)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) — lump in scrotum lipoma right neck cyst with discharge Left cheek papulae left kidney lesion on CT R elbow nodule/cyst
Nervous system disorders - Other, specify (Nervous system disorders) | 10 (12) — lightheadedness imbalances
Neutrophil count decreased (Investigations) | 16 (19)
Non-cardiac chest pain (General disorders) | 1 (1)
oral cavity fistula (Gastrointestinal disorders) | 6 (6)
Oral dysesthesia (Gastrointestinal disorders) | 6 (6)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 34 (43)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (General disorders) | 27 (31)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (18)
Papulopustular rash (Infections and infestations) | 2 (2)
Paresthesia (Nervous system disorders) | 16 (17)
Periodontal disease (Gastrointestinal disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 3 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (4)
Pharyngeal fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Phlebitis (Vascular disorders) | 1 (1)
photophobia (Eye disorders) | 1 (1)
Platelet count decreased (Investigations) | 13 (17)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Prostatic pain (Reproductive system and breast disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (7)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 2 (2) — ETOH cognitive dysfunction post-traumatic stress disorder
Psychosis (Psychiatric disorders) | 1 (1)
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 9 (11)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 11 (13)
Rash pustular (Infections and infestations) | 1 (1)
rectal pain (Gastrointestinal disorders) | 2 (2)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 3 (3) — dysuria nocturia nitrites, bacteria, and WBC in urine
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 12 (21) — Increased mucus rhonchi velopharyngeal inefficiency Subcutaneous emphysema
Salivary duct inflammation (Gastrointestinal disorders) | 14 (14)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1)
seroma (Injury, poisoning and procedural complications) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 12 (14)
Sinusitis (Infections and infestations) | 2 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 18 (19) — angular stomatitis oropharyngeal erythema skin breakdown posterior oropharynx erythema erythema cracked and bleeding lips Dermatitis Cellulitis autoimmune dermatitis Right facial skin blisters
skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
skin induration (Skin and subcutaneous tissue disorders) | 1 (1)
Skin infection (Infections and infestations) | 7 (7)
Skin ulceration (Skin and subcutaneous tissue disorders) | 4 (5)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Soft tissue infection (Infections and infestations) | 2 (2)
Somnolence (Nervous system disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 27 (37)
stomach pain (Gastrointestinal disorders) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 3 (3)
suicidal ideation (Psychiatric disorders) | 2 (2)
Superficial soft tissue fibrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Superficial thrombophlebitis (Vascular disorders) | 1 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Surgical and Medical Procedure - Other, specify (Surgical and medical procedures) | 8 (8) — total thyroidectomy and surgical dissection debulking flap intraoperative anastomosis failure Gastrostomy tube replacement Free Flap Failure
Syncope (Nervous system disorders) | 3 (3)
Thromboembolic event (Vascular disorders) | 3 (3)
Tinnitus (Ear and labyrinth disorders) | 15 (16)
Toothache (Gastrointestinal disorders) | 2 (2)
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tracheal obstruction (Injury, poisoning and procedural complications) | 1 (1)
Trigeminal nerve disorder (Nervous system disorders) | 1 (1)
Trismus (Musculoskeletal and connective tissue disorders) | 20 (24)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 3 (3)
Urinary retention (Renal and urinary disorders) | 3 (3)
Urinary tract infection (Infections and infestations) | 5 (8)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Vasovagal reaction (Nervous system disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 11 (12)
Vomiting (Gastrointestinal disorders) | 21 (30)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 48 (110)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (4)
White blood cell decreased (Investigations) | 13 (18)
Wound complication (Injury, poisoning and procedural complications) | 8 (10)
Wound dehiscence (Injury, poisoning and procedural complications) | 9 (11)
Wound Infection (Infections and infestations) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication but has the right to delay or extend publication or presentation timeframes for a period not to exceed 60 days after the initial review period when this would impact sponsor's ability to obtain patent protection.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/93/NCT02641093/Prot_SAP_000.pdf